CLINICAL TRIAL: NCT03486132
Title: Continuous Versus Interrupted Suturing In Repair of Lateral And Mediolateral Episiotomy
Brief Title: Repair of Lateral And Mediolateral Episiotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohammed mahmoud samy, Dr. Mohamed Samy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPI
Record Dates: First submitted 2016-04-25; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Episiotomy Wound

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- interrupted repair of mediolateral episiotomy (Other): using the interrupted suture (IT) which involves placing three layers of sutures: a continuous non-locking stitch to close the vaginal epithelium. commencing above the apex of the wound and finishing at the level of the fourchette; three or four interrupted sutures to reapproximate the deep and superficial perineal muscles; and interrupted transcutaneous technique to close the skin.
  The standard suture material in the study will be EGYSORB (sterile coated synthetic polyglycolic acid absorbable braided suture) No 2/0 Mediolateral episiotomy:it is defined as an incision beginning in the midline and directed laterally and downwards away from the rectum .The incision is usually about four centimeters long. In addition to the skin and subcutaneous tissues the bulbocavernosus, transverse perineal, and puborectalis muscles will be cut
  Interventions: Procedure: repair of episiotomy
- continous repair of mediolateral episiotomy (Other): continuous knotless suturing technique (CKT) which involves placing the first stitch above the apex of vaginal trauma to secure any bleeding points that might not be visible. Vaginal wound, perineal muscles (deep and superficial), and skin are reapproximated with a loose, continuous, non-locking technique. The skin sutures will be placed closely fairly deeply in the subcutaneous tissue, reversing back and finishing with a terminal knot placed in the vagina beyond the hymeneal remnants Mediolateral episiotomy:it is defined as an incision beginning in the midline and directed laterally and downwards away from the rectum .The incision is usually about four centimeters long. In addition to the skin and subcutaneous tissues the bulbocavernosus, transverse perineal, and puborectalis muscles will be cut The standard suture material in the study will be EGYSORB (sterile coated synthetic polyglycolic acid absorbable braided suture) No 2/0
  Interventions: Procedure: repair of episiotomy
- interrupted repair of lateral episiotomy (Other): using the interrupted suture (IT) which involves placing three layers of sutures: a continuous non-locking stitch to close the vaginal epithelium. commencing above the apex of the wound and finishing at the level of the fourchette; three or four interrupted sutures to reapproximate the deep and superficial perineal muscles; and interrupted transcutaneous technique to close the skin.
  The standard suture material in the study will be EGYSORB (sterile coated synthetic polyglycolic acid absorbable braided suture) No 2/0 And Lateral episiotomy; It begins in the vaginal introitus 1 or 2 cm lateral to the midline and is directe downwards towards the ischial tuberosity
  Interventions: Procedure: repair of episiotomy
- continuous repair of lateral episiotomy (Other): continuous knotless suturing technique (CKT) which involves placing the first stitch above the apex of vaginal trauma to secure any bleeding points that might not be visible. Vaginal wound, perineal muscles (deep and superficial), and skin are reapproximated with a loose, continuous, non-locking technique. The skin sutures will be placed closely fairly deeply in the subcutaneous tissue, reversing back and finishing with a terminal knot placed in the vagina beyond the hymeneal remnants And Lateral episiotomy; It begins in the vaginal introitus 1 or 2 cm lateral to the midline and is directe downwards towards the ischial tuberosity The standard suture material in the study will be EGYSORB (sterile coated synthetic polyglycolic acid absorbable braided suture) No 2/0
  Interventions: Procedure: repair of episiotomy

INTERVENTIONS:
Procedure: repair of episiotomy — Different techniques for repair of episiotomy incsicion

SUMMARY:
Episiotomy is an incision in the perineum carried out during the second stage of labour to facilitate the birth of an infant. It is an important surgical procedure with physiological, psychological and socio-economic effects on women. Therefore, not only the decision to carry out an episiotomy but also how it is performed and the quality of aftercare are important The two most often performed are the lateral and median episiotomy, as well as mediolateral episiotomy.

Two common methods of repair of episiotomy include continuous and interrupted methods This study aims to compare between postoperative pain following repair of episiotomy by continuous or interrupted suturing.

DETAILED DESCRIPTION:
Aim of the work:

This study aims to compare between postoperative pain following repair of episiotomy by continuous or interrupted suturing.

Study population:

All primipara full term women with episiotomy done in a selective rather than liberal use.

E- Patients in the study will be randomized into one of two groups either those who have:

1. Interrupted technique of episiotomy repair or
2. Continuous knotless suturing technique and each of the two groups will be subdivided into either medio-lateral or lateral episiotomy.

The Episiotomy in group A will be done using the interrupted suture (IT) which involves placing three layers of sutures: a continuous non-locking stitch to close the vaginal epithelium. commencing above the apex of the wound and finishing at the level of the fourchette; three or four interrupted sutures to reapproximate the deep and superficial perineal muscles; and interrupted transcutaneous technique to close the skin.

The Episiotomy in group B will be done using the continuous knotless suturing technique (CKT) which involves placing the first stitch above the apex of vaginal trauma to secure any bleeding points that might not be visible. Vaginal wound, perineal muscles (deep and superficial), and skin are reapproximated with a loose, continuous, non-locking technique. The skin sutures will be placed closely fairly deeply in the subcutaneous tissue, reversing back and finishing with a terminal knot placed in the vagina beyond the hymeneal remnants.

And subgroups subjected to Mediolateral episiotomy:it is defined as an incision beginning in the midline and directed laterally and downwards away from the rectum .The incision is usually about four centimeters long. In addition to the skin and subcutaneous tissues the bulbocavernosus, transverse perineal, and puborectalis muscles will be cut. And Lateral episiotomy; It begins in the vaginal introitus 1 or 2 cm lateral to the midline and is directe downwards towards the ischial tuberosity.

The standard suture material in the study will be EGYSORB (sterile coated synthetic polyglycolic acid absorbable braided suture) No 2/0, Manufacturer TAISIER-MED Company).

F- Written informed consent will be taken from all women participating in our search.

G- Data recording: age,weight,height,body mass index,type of anesthesia used,type of episiotomy,time taken,infection or gaped episiotomy, amount of bleeding, postpartum hemorrhage,amount of suture material used,amount of analgesia used, severity of pain detected by VAS.

H- all patient will be given oral nonnarcotic analgesics (NSAIDs eg; ibuprofen 600 mg every eight hours for three days , if NSAIDs is contraindicated acetaminophen/ paracetamol 500 mg every eight hours for three days.

I- Antibiotic prophylaxis will be given as a single dose of a broad spectrum antibiotic (second generation cephalosporin or clindamycin if the patient is allergic to penicillin

ELIGIBILITY:
Inclusion criteria:

1. Primipara women.
2. Fullterm pregnancy.
3. Lateral or mediolateral episiotomy done in selective rather than liberal episiotomy.

Exclusion Criteria:

1. Risk factor of trauma eg; macrosomia, congenital fetal malformations as (exophthalmous major, hydrocephalus, spinal cord teratoma….etc.
2. Instrumental delivery.
3. Primipara refuses to be in the study.
4. Other techniques of episiotomy.
5. Preterm onset of labour.
6. Indication for CS eg; CPD, malposition and malpresentation, fetal distress….etc.
7. Use of epidural analgesics.
8. Factors affecting wound healing eg;DM, corticosteroid therapy, chronic debilitating diseases…etc.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 6 hours
  using visual analogue scale

SECONDARY OUTCOMES:
Postoperative pain two monthes after delivery. | TWO MONTHS
  using VAS
Time taken in repair (min) | 1 hour
Number of suture ampoules used. | 1 hour
Dyspareunia | two months
  Dyspareunia reported up to two months after delivery (ACOG;1995). according to Marinoff dyspareunia scale:
  0 = no dyspareunia;
  1. = causes discomfort, but does not interfere with the frequency of intercourse;
  2. = sometimes prevents intercourse; and
  3. = completely prevents intercourse.
Early complication of episiotomy eg; anal spincter injury, rectal mucosal injury, bleeding or heamatoma formation. | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No